CLINICAL TRIAL: NCT02656121
Title: Correction of Vitamin D Deficiency and Its Effect on Ovulation Induction in Women With PCOS (VIDEO): A Feasibility RCT
Acronym: PCOSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed El Kotb Abdel Fattah, Dr. Ahmed Kotb, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCO
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: PCOS
Keywords: PCOS, vitamin D
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Vitamin D; Clomiphene; Ovulation Induction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Experimental): 1st subgroup will be tested and treated with vitamin D together with Clomiphene Citrate for induction of ovulation
  Interventions: Drug: Vitamin D; Drug: Ovulatory Agent
- control (Active Comparator): 2nd subgroup will be treated with Clomophene Citrate only
  Interventions: Drug: Ovulatory Agent

INTERVENTIONS:
Drug: Vitamin D — 6000 IU of vitamin D3
  Other Names: Vidrop®, Medical Union Pharmaceuticals, Egypt
  Arms: Vitamin D
Drug: Ovulatory Agent — only Clomophine Citrate
  Other Names: Clomiphene Citrate for induction of ovulation

SUMMARY:
Recently, a special emphasis has recently been directed to the potential role of vitamin D and some regulatory peptides (e.g. adipokines and follistatin) and their associated metabolic roles and genetic factors in the development of PCOS and its related co-morbidities. The aim of this study was to assess the feasibility of conducting a pragmatic RCT assessing the effectiveness of adopting a protocol of screening for and correcting Vitamin D deficiency in women with PCOS seeking fertility treatment in a low/middle income care (LMIC) setting

DETAILED DESCRIPTION:
Research question:

In PCOS patients, is there any effect of vitamin D testing and correction on ovulation induction in women with PCOS?

Research hypothesis:

There is effect of testing and correcting vitamin D status as regard ovulation in patients with PCOS

ELIGIBILITY:
Inclusion Criteria:

* diagnosed PCOS cases according to the National Institute of Health criteria (NIH consensus criteria) and Rotterdam criteria

Exclusion Criteria:

* 1- PCOS patients not in child bearing age; less than 18 years or more than 45 years.

  2- Patients with congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome, hyperprolactinemia and virilizing ovarian or adrenal tumors.

  3- PCOS patients with any other medical illness. 4- PCOS patients already on vitamin D supplements.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
cumulative clomiphene citrate-induced ovulation rates | 6 months
  Ultrasound Folliculometry was performed every other day starting on the 10th day of the induction cycle. Until, at least, one follicle reached 18mm in diameter

SECONDARY OUTCOMES:
Cumlative clinical pregnancy rate | 6 months
  detection of fetal heart activity detected by transvaginal ultrasound
median ovulating dose of clomiphene citrate | 6 months
  Dose required

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M kotb, MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes